CLINICAL TRIAL: NCT03415555
Title: Efficacy of Erector Spinae Plane (ESP) Blockade in Patients Scheduled for Minimally Invasively Mitral Valve Replacement
Brief Title: Postoperative Analgesia After Minithoracotomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Lublin (Other)
Collaborators: University of Rzeszow (Other)
Responsible Party: Principal Investigator, Michał Borys, associate professor, Medical University of Lublin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KE-0254/26/2018
Record Dates: First submitted 2018-01-23; First posted 2018-01-30 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Postoperative Pain; Mitral Valve Disease
Keywords: Erector Spinae Plane blockade; patient control anlagesia; mitral valve replacement
MeSH Terms: conditions — Pain, Postoperative | interventions — Oxycodone; Passive Cutaneous Anaphylaxis; Anesthesia, General; Acetaminophen

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant
Masking Description: Single (Participant)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESP (Experimental): Before the induction of general anesthesia, Erector Spinae Plane (ESP) blockade will be done. Postoperative analgesia is provided with intravenous oxycodone. Patient-controlled analgesia pump (PCA) will be used for this purpose.
  Interventions: Procedure: Erector Spinae Plane blockade; Drug: Oxycodone; Procedure: general anesthesia; Drug: paracetamol
- PCA (Experimental): Postoperative analgesia is provided with intravenous oxycodone. Patient-controlled analgesia pump (PCA) will be used for this purpose. ESP will not be done in this arm.
  Interventions: Drug: Oxycodone; Procedure: general anesthesia; Drug: paracetamol

INTERVENTIONS:
Procedure: Erector Spinae Plane blockade — Before the beginning of the procedure, ESP blockade will be performed under ultrasound control. A single-shot technique will be used with 0.375 % solution of ropivacaine: 0.2 mL per patients' KG. The maximum dose is 40 mL.
  Other Names: ESP
  Arms: ESP
Drug: Oxycodone — Each patient, before the end of surgery, will be administered i.v. 0.1 mg of oxycodone. PCA with oxycodone (1mg/mL) will be utilized during the postoperative period: 5-minute interval.
  Other Names: PCA with oxycodone
Procedure: general anesthesia — Each patient will generally anesthetized and endotracheal tube will be inserted
  Other Names: GA
Drug: paracetamol — Paracetamol will be given i.v. every 6 hours.

SUMMARY:
Patients scheduled for minimally invasive mitral valve replacement. Each patient will be treated with intravenous (i.v.) oxycodone - patient-controlled analgesia (PCA). Half of the patients will be randomly allocated to Erector Spinae Plane (ESP) blockade group.

DETAILED DESCRIPTION:
Only patients who are qualified for an elective procedure of mitral valve replacement may participate in the study. Each patient will be anesthetized generally. The same drugs will be used in each stage of anesthesia. The induction: etomidate, remifentanil, rocuronium, scolina as required. The maintenance: sevoflurane, remifentanil, rocuronium. The emergence: oxygen, sugammadex or neostigmine a required.

Patients will be randomly allocated into one of two groups: PCA or ESP. Among the patients from ESP group will have ESP blockade before the induction of general anesthesia. ESP blockade will be performed under ultrasound control. A single-shot technique will be used with 0.375 % solution of ropivacaine: 0.2 mL per patients' KG. The maximum dose is 40 mL.

Each patient, before the end of surgery, will be administered i.v. 0.1 mg of oxycodone. PCA with oxycodone (1mg/mL) will be utilized during the postoperative period: 5-minute interval. This is standard protocol in our department.

Only patients who are successfully awakened after the procedure may participate in the study.

The pain intensity will be assessed with visual-analogue scale (VAS) at 2, 4, 8, 12 and 24 hour after the end of anesthesia.

The total consumption of oxycodone will be also monitored.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled mitral valve replacement surgery
* obtained consent

Exclusion Criteria:

* allergy to oxycodone and local anesthetics
* depression, antidepressant drugs treatment
* epilepsy
* usage of painkiller before surgery
* addiction to alcohol or recreational drugs
* postoperative ventilation or ICU admission

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-02-07 (Actual); Primary Completion 2018-04-18 (Actual); Study Completion 2018-04-18 (Actual)

PRIMARY OUTCOMES:
Pain intensity | From the end of anesthesia till 24 hour postoperatively. VAS range from 0 (no pain, good outcome) to 100 in millimeters (the worst pain ever, bad outcome).
  Patients' self-pain assessment with VAS (visual-analogue scale)

SECONDARY OUTCOMES:
Total consumption of oxycodone | From the end of anesthesia till 24 hour postoperatively
  The cumulative consumption of oxycodone during 24 hour from the end of anesthesia.

CONTACTS AND LOCATIONS:
Overall Officials: Mirosław Czuczwar, M.D., PhD, Study Chair — Medical University of Lublin
Locations (1):
- Queen Jadwiga Hospital, Rzeszów, Poland